CLINICAL TRIAL: NCT05406232
Title: Quantifying Temporal Immunologic Changes With Hypofractionated Radiation-Induced DNA Damage in Breast Cancer
Brief Title: Temporal Immunologic Changes With Hypofractionated Radiation-Induced DNA Damage in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Artidis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-0669; NCI-2021-09773 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0669 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma; Invasive Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; Radiotherapy; Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (RT, biopsy): Patients undergo RT on day 1. Patients also undergo tumor punch biopsies and blood sample collection prior to the first fraction and on days 1, 3, and 7.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor punch biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This study assesses changes to the immune cells following hypofractionated radiation-induced DNA damage in breast cancer patients. Radiation therapy may cause immune cells to enter tumors and target cancer cells. The goal of this study is to measure the change in the level of immune cells in the tumor before and after radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the percent change in immune infiltration at day 3 and day 7 of radiotherapy (RT) relative to baseline (before radiotherapy).

SECONDARY OBJECTIVE:

I. To estimate the degree of deoxyribonucleic acid (DNA) damage at approximately 3 and 7 days after radiotherapy compared to baseline.

II. To examine cancer cell intrinsic immune signaling following radiotherapy.

EXPLORATORY OBJECTIVE:

I. To examine the association between DNA damage and micronuclei formation. II. To examine the association between DNA damage and immune infiltration. III. To examine the association between micronuclei formation and immune infiltration.

OUTLINE:

Patients undergo RT on day 1. Patients also undergo tumor punch biopsies and blood sample collection prior to the first fraction and on days 1, 3, and 7.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age with biopsy proven invasive breast cancer
* Breast cancer that appears to be superficially accessible to a tumor punch biopsy
* Patients thought to derive clinical benefit from palliative RT to the breast/chestwall
* In discussions with the medical oncologist, if clinically reasonable, systemic therapy will be held during RT

Exclusion Criteria:

* A history of prior radiation to the area requiring radiation for which the attending physician believes reirradiation could not be safely delivered
* Pregnancy
* Active usage of anticoagulant medications that are considered to pose an increased risk of tumor punch biopsies
* Receipt of immunotherapy or chemotherapy 7 days prior to start of RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer that appears to be superficially accessible to a tumor punch biopsy
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To estimate the percent change in immune infiltration. | Baseline up to day 7
  Will be estimated with corresponding two-sided 80% confidence intervals. Also, marker levels at each time point and unstandardized effect sizes (arithmetic differences from baseline) across time points will be estimated along with 2-sided 80% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Simona F Shaitelman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org